CLINICAL TRIAL: NCT05052528
Title: A Phase I Study to Evaluate the Safety of Escalating Doses of Lymphodepleting Conditioning Chemotherapy Prior to CD19 Chimeric Antigen Receptor T Cells in Subjects With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Fludarabine and Cyclophosphamide With or Without Rituximab Before CD19 Chimeric Antigen Receptor T Cells for the Treatment of Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mehrdad Abedi, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mehrdad Abedi, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#299; NCI-2021-07396 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#299 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Immunotherapy, Adoptive; Cyclophosphamide; fludarabine phosphate; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose level 1 (fludarabine, cyclophosphamide, CD19 CAR T) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes daily and cyclophosphamide IV over 60 minutes daily on days -5 to -3. Patients also receive CD19 CAR T cells IV on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate
- Dose level 2 (rituximab, fludarabine, cyclophosphamide, CAR T) (Experimental): Patients receive rituximab IV on day -5, fludarabine phosphate IV over 30 minutes daily on days -5 to -3, and cyclophosphamide IV over 60 minutes on days -5 to -3. Patients also receive CD19 CAR T cells IV on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Biological: Rituximab
- Dose level 3 (fludarabine, cyclophosphamide, CD19 CAR T) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes daily on days -3 to -5 and cyclophosphamide IV over 60 minutes daily on day -5. Patients also receive CD19 CAR T cells IV on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate
- Dose level 4 (rituximab, fludarabine, cyclophosphamide, CAR T) (Experimental): Patients receive rituximab IV on day -5, fludarabine phosphate IV over 30 minutes daily on days -5 to -3, and cyclophosphamide IV over 60 minutes on day -5. Patients also receive CD19 CAR T cells IV on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Biological: Rituximab
- Dose level 5 (fludarabine, cyclophosphamide, CD19 CAR T) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes daily on days -5 to -1 and cyclophosphamide IV over 60 minutes daily on days -5 and -4. Patients also receive CD19 CAR T cells IV on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate
- Dose level 6 (rituximab, fludarabine, cyclophosphamide, CAR T) (Experimental): Patients receive rituximab IV on day -5, fludarabine phosphate IV over 30 minutes daily on days -5 to -1, and cyclophosphamide IV over 60 minutes on days -5 and -4. Patients also receive CD19 CAR T cells IV on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Biological: Rituximab

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given CD19 CAR T cells IV
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
  Arms: Dose level 2 (rituximab, fludarabine, cyclophosphamide, CAR T); Dose level 4 (rituximab, fludarabine, cyclophosphamide, CAR T); Dose level 6 (rituximab, fludarabine, cyclophosphamide, CAR T)

SUMMARY:
This phase I trial evaluates the best dose, possible benefits and/or side effects of fludarabine and cyclophosphamide with or without rituximab before CD19 chimeric antigen receptor T cells in treating patients with diffuse large B-cell lymphoma that has come back (relapsed) or has not responded to previous treatment (refractory). T-cells are a normal part of the immune system. To make the T-cell medication, T-cells are taken from the blood and altered in a laboratory. They are then returned to the body. The altered T-cells will latch on to a specific part of the cancer cells and hopefully kill them. Once the T-cells have been altered in the laboratory, they are called "CAR T-cells." CAR is short for "chimeric antigen receptors." These are structures on the surface of cells that allow the altered T-Cells to find and destroy the cancer cells. Another part of the T-Cell medication is called "CD19." This part is called a "biomarker." Biomarkers help doctors determine whether a cancer is getting worse and whether medications are working to stop it. The chemotherapy drugs that are given before the T-Cell therapy are cyclophosphamide, fludarabine and rituximab. Rituximab is an immunotherapy drug. These chemotherapy drugs will reduce the number of normal (unaltered) T-Cells in the body to make room for the altered T-cells to kill the cancer cells. Giving fludarabine and cyclophosphamide with or without rituximab before CD19 CAR T cell therapy may help improve response to CD19 CAR T cell therapy in patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:I. To examine the feasibility to manufacture autologous CD19 CAR T cells at a minimum target dose of 1.0 x 10^6 cells/kilogram using the CliniMACS automated system.II. To determine the safety of administering high-dose conditioning chemotherapy with cyclophosphamide and fludarabine with rituximab prior to CD19 CAR-T cell therapy in patients with relapsed (R)/refractory (R) diffuse large B cell lymphoma (DLBCL) and to find the recommended regimen after phase II dose for this therapy.III. To determine the safety of infusion of chimeric antigen receptor T cells targeting CD19 in adults with R/R DLBCL.

SECONDARY OBJECTIVES:I. To describe the toxicities related to CD19 targeted CAR T cells.II. To describe the overall response rate (ORR) and complete response (CR) rate of relapsed DLBCL treated with CD19 CAR T cells.III. To assess other response variables including overall survival (OS), progression free survival (PFS), and event free survival (EFS).

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 6 dose levels.

DOSE LEVEL 1: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes daily and cyclophosphamide IV over 60 minutes daily on days -5 to -3. Patients also receive CD19 CAR T cells IV on day 0.

DOSE LEVEL 2: Patients receive rituximab IV on day -5, fludarabine phosphate IV over 30 minutes daily on days -5 to -3, and cyclophosphamide IV over 60 minutes on days -5 to -3. Patients also receive CD19 CAR T cells IV on day 0.

DOSE LEVEL 3: Patients receive fludarabine phosphate IV over 30 minutes daily on days -3 to -5 and cyclophosphamide IV over 60 minutes daily on day -5. Patients also receive CD19 CAR T cells IV on day 0.DOSE LEVEL 4: Patients receive rituximab IV on day -5, fludarabine phosphate IV over 30 minutes daily on days -5 to -3, and cyclophosphamide IV over 60 minutes on day -5. Patients also receive CD19 CAR T cells IV on day 0.

DOSE LEVEL 5: Patients receive fludarabine phosphate IV over 30 minutes daily on days -5 to -1 and cyclophosphamide IV over 60 minutes daily on days -5 and -4. Patients also receive CD19 CAR T cells IV on day 0.

DOSE LEVEL 6: Patients receive rituximab IV on day -5, fludarabine phosphate IV over 30 minutes daily on days -5 to -1, and cyclophosphamide IV over 60 minutes on days -5 and -4. Patients also receive CD19 CAR T cells IV on day 0.After completion of study treatment, patients are followed up at 30, 60, and 90 days, 6 and 12 months, and then annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Commercial CD19 CAR T cell product not available for the patient
* Male or female, aged >= 18
* In good general health as evidenced by medical history or as determined by the principal investigator (PI)
* Ability to swallow oral medication and willingness to adhere to the study intervention and any required medications
* For females of reproductive potential: use of highly effective contraception (oral contraceptives, intrauterine device) during screening confirmed with serum pregnancy test, and agreement to use such a method during study participation and for an additional 4 weeks after the end of CD19 CAR T cell infusion
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
* Agreement to adhere to lifestyle considerations throughout study duration including abstaining from tobacco and drug use
* Subjects must have relapsed or refractory diffuse large B cell lymphoma treated with at least two lines of therapy Subjects must have failed to have a complete response, or have recurrent disease after the last treatment regimen. Subjects must have previously been treated with a regimen that includes an anthracycline and an anti-CD20 monoclonal antibody. Autologous transplant will be counted as one line of therapy
* The patient's disease must be CD19 positive, either by immunohistochemistry or flow cytometry analysis on the last biopsy available
* Age >= 18 years
* Performance status: Adult Subjects: Eastern Cooperative Oncology Group (ECOG) >= 1; Subjects > 10 years of age: Karnofsky >= 80%
* Absolute neutrophil count (ANC) >= 1000
* Platelets >= 100/mm^3
* Hemoglobin > 8 g/dL
* ANC >= 500 is acceptable if documented bone marrow involvement by disease
* Creatinine clearance (estimated by Cockcroft Gault) or using 24 hour (hr) urine collection >= 50 cc/min
* Total bilirubin =< 2 mg/dL except in subjects with Gilbert's Syndrome in whom total bilirubin must be =< 3.0
* Alanine transaminase (alanine aminotransferase [ALT]/serum glutamic pyruvic transaminase [SGPT]) and aspartate aminotransferase (aspartate aminotransferase [AST]/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x the upper limit of normal or =< 5 x the upper limit of normal if documented liver involvement by disease
* Cardiac left ventricular ejection fraction >= 45% as determined by an echocardiogram and no clinically significant electrocardiogram (ECG) findings
* Baseline oxygen saturation > 92% on room air
* Prior cancer directed therapy wash-out: at least 2 weeks or 5 half-lives, whichever is shorter must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for radiotherapy within 10 days of apheresis, systemic corticosteroid use within 7 days of apheresis (with the exception of single dose for an allergic reaction), or any other immunosuppressive therapies within 7 days
* No use of lymphodepleting agents including alemtuzumab and antithymocyte globulin for 7 days prior to peripheral blood collection, 5 days prior to CD19 CAR T cell infusion and for 90 days after infusion

Exclusion Criteria:

* Presence of supplemental oxygen, cardiac pacemaker
* Known allergic reactions to components of the anti-CD19 CAR T cell product as evidenced by prior documented anaphylactic reaction or other clinical signs and/or symptoms of an allergic reaction as determined by the PI
* Febrile illness within 3 days of admission for lymphodepleting conditioning therapy
* Treatment with another investigational drug or other investigational intervention within 2 weeks of apheresis
* Primary immunodeficiency
* History of autoimmune diseases (ex: Crohn's, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's) resulting in end organ damage or requiring systemic immunosuppressive or systemic disease modifying agents within the last two years prior to enrollment
* Autologous transplant within 6 weeks and allogeneic transplant within 3 months of planned CAR T cell infusion
* Recipient of CD19 CAR T cell therapy outside of this protocol
* Active central nervous system or meningeal involvement by tumor. Subjects with untreated brain metastases/central nervous system (CNS) disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal involvement must be in a documented remission by cerebrospinal fluid (CSF) evaluation and contrast-enhanced magnetic resonance imaging (MRI) for at least 30 days prior to study enrollment
* History of active malignancy other than non-melanoma skin cancer, carcinoma in situ (e.g. cervix, bladder, breast)
* Active human immunodeficiency virus (HIV) infection documented by positive viral load
* Subjects with uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study because CAR T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four (4) weeks after receiving the CAR-T cell infusion
* Diagnosis of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of products successfully manufactured meeting the established release criteria with a goal of at least 1.0 x 10^6 cells/kilogram | Up to 15 years
Incidence and severity of adverse events related to lymphodepleting chemotherapy and or CD19 chimeric antigen receptor (CAR) T cells | 2 months
  Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate and the toxicity rate. Toxicity data by type and severity will be summarized by frequency tables.
Dose limiting toxicities (DLTs) related to lymphodepleting chemotherapy and or CD19 CAR T cells | 2 months
  Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate and the toxicity rate. Toxicity data by type and severity will be summarized by frequency tables.
Maximum tolerated dose | 2 months
Incidence and severity of DLT associated with infusion of CD19 CAR T cells (infusion reactions) | 2 months
  Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate and the toxicity rate. Toxicity data by type and severity will be summarized by frequency tables.

SECONDARY OUTCOMES:
Incidence of toxicities related to CD19 CAR T cells | Up to 15 years
  Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate and the toxicity rate. Toxicity data by type and severity will be summarized by frequency tables.
Overall response rate | At 3 months after completion of CAR-T therapy
  Defined as the percentage of patients that achieve partial response or complete response. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate and the toxicity rate.
Complete response rate | At 3 months after completion of CAR T therapy
  Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate and the toxicity rate.
Overall survival | From the start of the conditioning lymphodepletion chemotherapy on day -6 until death, assessed at 1 year
  Will be estimated using Kaplan and Meier methods. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Progression free survival | From the start of the conditioning lymphodepletion chemotherapy regimen until the documentation of disease progression or death due to any cause, whichever occurs first, assessed at 1 year
  Will be estimated using Kaplan and Meier methods. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Event free survival | From the date of day -6 of lymphodepleting conditioning therapy to the date of first documented progression, initiation of new anti-lymphoma treatment, or death, assessed at 1 year
  Will be estimated using Kaplan and Meier methods. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Abedi, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States